CLINICAL TRIAL: NCT05430711
Title: Induction of Labour With Dinoprostone vs. Expectant Management After Prelabour Rupture of Membranes at Term
Brief Title: Dinoprostone Induction vs. Expectant Management After PROM at Term
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Polona Peclin, Principal investigator, University Medical Centre Ljubljana
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0120-115/2019/13
Record Dates: First submitted 2022-06-11; First posted 2022-06-24 (Actual); Last update posted 2022-06-24 (Actual); Status verified 2022-06

CONDITIONS: Prelabor Rupture of Membranes
Keywords: Induction of labour; Dinoprostone; Cervical ripening
MeSH Terms: conditions — Fetal Membranes, Premature Rupture | interventions — Dinoprostone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dinoprostone (Experimental): Participants will receive dinoprostone 10 mg vaginal delivery system for up to 24 hours.
  Interventions: Drug: Dinoprostone
- Expectant management (No Intervention): Participants will not receive drugs to induce labour, they will be managed expectantly for up to 24 hours.

INTERVENTIONS:
Drug: Dinoprostone — After randomization, participants will receive dinoprostone 10 mg vaginal delivery system which will remain in place up to 24 hours or until the labour begins. At the onset of labor or after 24h it will be removed and participant transferred to labour room for further standard procedures.
  Other Names: Propess
  Arms: Dinoprostone

SUMMARY:
Prelabour rupture of membranes (PROM) is associated with intrauterine infection and maternal and neonatal consequences. This risk increases with the length of time from PROM to delivery. Induction of labor has been shown to reduce the rates of those complications, however the optimal time interval has not yet been determined.

The main purpose of this single-center randomized prospective study is to assess the differences between two approaches of managing PROM at term-expectant management and induction with a dinoprostone vaginal delivery system.

DETAILED DESCRIPTION:
Women with singleton pregnancy in cephalic presentation at term (37-41 6/7 weeks gestational age) will be randomised 4 to 12 hours after PROM when a sterile vaginal exam will be completed to assign Bishop score. When Bishop score at presentation will be ≤5, the study will be presented to the patient. Once the patient will be consented and randomized, women will receive dinoprostone vaginal delivery system (for up to 24 hours after randomisation) or will be managed expectantly (for up to 24 hours after randomisation).

Patients randomized to the expectant management group will be admitted to the maternity ward, where they will wait up to a maximum of 24 hours for labor to start spontaneously.

Patients in the induction group will also be admitted to the maternity ward and induced with a dinoprostone vaginal delivery system. If not removed sooner, the vaginal delivery system will be removed after 24h.

If patients in both groups will not be in active labor 24 hours after randomisation they will be admitted to the delivery room and health care providers will manage active labor per usual practice. The need for cesarean section or operative delivery or will be at the discretion of the healthcare provider.

In the days following birth, woman in both groups, will be asked to fill in a questionnaire about their satisfaction with the labour experience.

ELIGIBILITY:
Inclusion Criteria:

* 4 to12 hours after prelabour rupture of membranes
* 18-50 years of age
* Parity 0 to 2
* Singleton pregnancy
* Cephalic presentation
* Term (37-41 6/7 weeks gestational age)
* Bishop score ≤5
* Reassuring fetal status

Exclusion Criteria:

* Uterine contractions
* Signs of infection
* Signs of non-reassuring fetal status
* Meconium-stained amniotic fluid
* Group B Streptococcus colonization
* Fetal demise or major congenital anomaly
* Intrauterine growth restriction (estimated fetal weight ≤ 3 percentile)
* Contraindications for vaginal birth or use of prostaglandins for labor induction

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Pregnant women
Enrollment: 70 (Estimated)
Dates: Start 2022-06 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Time from randomisation to delivery | Within 1 week
  Time measured from randomisation to the delivery time

SECONDARY OUTCOMES:
Time from randomisation to spontaneous vaginal delivery | Within 1 week
  Time measured from randomisation to the spontaneous vaginal delivery (delivery without the use of forceps, vacuum extraction, or a cesarean section)
Time from PROM to delivery | Within 1 week
  Time measured from prelabor rupture of membrane (leaking of amniotic fluid) until delivery
Cesarean delivery rate | Within 1 week
  Percentage of patients who deliver via cesarean section for whatever reason
Instrumental delivery rate | Within 1 week
  Percentage of patients who deliver via instrumental delivery (forceps, a vacuum device) for whatever reason
Use of oxytocin | Within 1 week
  Oxytocin used prior to the delivery of the baby. If oxytocin was used, we will measure how many international units (IU) of oxytocin were used from the beginning of labor to the delivery of the baby.
Hyperstimulation with nonreassuring fetal heart rate tracing | Within 1 week
  Percentage of uterine hyperstimulation- exaggerated uterine response consisting of uterine hypertonus, a single uterine contraction lasting two or more minutes or uterine tachysystole with a least 12 contractions in 20 minutes, with a simultaneous nonreassuring fetal heart rate tracing as defined by the 2015 FIGO (The international federation of gynaecology and obstetrics) classification of intrapartum cardiotocography.
Rate of chorioamnionitis | Within 1 week
  Clinical chorioamnionitis (a fever of 38.0°C or more plus one or more of the following: baseline fetal heart rate > 160 beats/minute for ≥ 10 minutes, maternal white cell count >15,000 cells/mm3 or purulent-appearing fluid coming from the cervical os visualized by speculum examination).
Rate of endometritis | Within 3 weeks
  Clinical endometritis (postpartum woman with at least two of the following signs or symptoms: fever ≥38.0°C, pain or tenderness (uterine or abdominal) with no other recognized cause or purulent drainage from the uterus.)
Rate of postpartum maternal fever | Within 3 weeks
  A fever of 38.0°C or more in the postpartum period.
Use of antibiotics | Within 3 weeks
  Possible use of antibiotics in the postpartum period.The decision of the need of antibiotics in the postpartum period is in the discretion of the physician.
Lenght of antibiotic treatment | 3 weeks
  The decision of the need of antibiotics in the postpartum period is in the discretion of the physician. If antibiotics will be used, we will measure length of antibiotic treatment (in days).
Number of neonates, admitted to intensive care unit | Within 3 weeks
  Infants which will be admitted to the neonatal intensive unit for whatever reason.
APGAR scores | Within 1 week
  Infants with a 5-minute APGAR score of less than 7.The Apgar score is a number calculated by scoring the heart rate, respiratory effort, muscle tone, skin color, and reflex irritability of the infant, 5 min after birth. Each of these objective signs can receive 0, 1, or 2 points. The higher is the sum of the points, the better is the condition of the newborn.
Maternal Length of Stay | Within 3 weeks
  Total length of hospitalization of women in days.
Rate of early neonatal sepsis | Within 3 weeks
  Infants with early neonatal sepsis, a diagnosis based on a positive blood, cerebrospinal fluid, or urine microbiological culture in the first 72 hours after birth.
Patients perception of labor (length, pain, overall satisfaction) | Within 3 weeks
  Satisfaction and perceptions of woman giving birth with labour through a self-administered questionnaire that they will answer in the postpartum period (6 to 48 hours after labor). They will specify their level of agreement or disagreement on a symmetric 4-point agree-disagree scale (1- I strongly disagree, 2- I disagree, 3- I agree, 4- I strongly agree) for a series of statements regarding aspects of birth.
  With the beforementioned scale we will measure patients' perception of length of hospitalization before childbirth, perception of pain before admission to the labour room, pain associated with vaginal examinations and insertion of the vaginal insert and if they would choose the same method of managing birth in the next pregnancy.

IPD SHARING:
Plan to Share IPD: No
IPD will be available on request